CLINICAL TRIAL: NCT03799770
Title: Optic Nerve Sheath Diameter as A Predictor of Early Tacrolimus Neurotoxicity After Living Donor Liver Transplantation
Brief Title: ONSD and Neurotoxicity in Liver Transplant
Status: Completed | Type: Observational
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Amr M. Yassen, professor of anaesthesia and surgical intensive care, Mansoura University
Other Study IDs: R.18.12.369 - 2018/12/16
Record Dates: First submitted 2019-01-06; First posted 2019-01-10 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Liver Transplant; Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Optic nerve sheath diameter by ultrasound at 5 minutes post-reperfucion — Patients were placed in the supine position with their eyes closed, and a thick gel layer was applied to the closed upper eyelid. The 7.5-MHz linear probe was placed on the gel without excessive pressure and adjusted to the proper angle for displaying the entry of the optic nerve into the globe. The intensity of the ultrasound was adjusted to display optimal contrast between the retrobulbar echogenic fat tissue and the vertical hypoechoic band. An ultrasound beam was focused on the retrobulbar area using the lowest possible acoustic power that could measure ONSD. The ONSD was measured 3 mm behind the optic disc. Measurements were performed in the transverse and sagittal planes of both eyes, and the ﬁnal ONSD value was calculated by average 4 measured values.
  We measured the ONSD at 4 timings: (T1) Post induction and before surgical incision, (T2) Portal vein clamping, (T3) 5 minutes after reperfusion, and (T4) 30 min after reperfusion.

SUMMARY:
This is a diagnostic test accuracy study. The investigators measure optic nerve sheath diameter (ONSD) by ultrasound on the eye during living donor liver transplantation operation at 5 minutes after reperfusion to predict the occurrence of early tacrolimus neurotoxicity after liver transplantation.

We measured the ONSD at 4 timings: (T1) Post induction and before surgical incision, (T2) Portal vein clamping, (T3) 5 minutes after reperfusion, and (T4) 30 min after reperfusion.

DETAILED DESCRIPTION:
Neurotoxicity is mainly associated with tacrolimus and cyclosporin, amounting to 10 - 30% for CS and up to 32% for tacrolimus.(2) . Sirolimus, everolimus, and mycophenolate mofetil lack the neurotoxicity of calcineurin inhibitors (3-4).

Neurotoxicity mostly occurs in the early postoperative period increasing morbidity, mortality and hospital and intensive care stay. Neurotoxicity has variable manifestations and mainly affects the CNS. They are usually divided into minor manifestations as tremor, headache, insomnia and paraesthesia or major encephalopathy, akinetic mutism, seizures, speech disorders, polyneuropathy, myopathy, pseudobulbar palsy and even stroke. (2) The main pathogenesis of calcinurin inhibitors neurotoxicity appears to be ﬂuid extravasation (vasogenic edema) due to disruption of blood brain barrier, not cell destruction (cytotoxic edema).(5) During liver transplant operation there are changes in the intracranial pressure and cerebral perfusion pressure especially during reperfusion that may affect the integrity of blood brain barrier. (6) There are multiple methods for monitoring of intracranial pressure invasive or non -invasive. The invasive method remains the gold standard for monitoring of intracranial pressure but there is a controversy about its use in liver transplantation as it may be complicated by bleeding and infections (7).

Also there are a multiple non-invasive methods for monitoring of ICP. Ultrasonographic measurement of the optic nerve sheath diameter (ONSD) was introduced recently as a useful noninvasive method for evaluating ICP. ONSD demonstrated a good correlation with the ICP level in many previously published studies. (8,9) Rajajee et al. found that the optimal cutoff of ONSD for the detection of an acutely increased ICP > 20 mm Hg was greater than 4.8 mm. (10) We hypothesize that the absolute value or the changes of ONSD during different stages of living donor liver transplantation operation may predict occurrence of early calcinurin inhibitor neurotoxicity (CNIN).We will investigate whether the absolute value or changes of ONSD during different stages of living donor liver transplantation operation may be a predictor of early calcinurin inhibitor neurotoxicity in the first month post liver transplantation. This is a prospective observational cohort study that will be conducted to all adult patients of both sex undergoing living donor liver transplantation operation at Gastro-Intestinal Surgical Centre (GISC), Mansoura university Hospitals, Mansoura, Egypt over the period covering more than 100 consecutive cases. After Institutional review board approval, we will secure informed consents from all included patients during the preoperative visits.

Anesthesia and surgery techniques will be done according to our center's protocol.(11)

Reperfusion:

On portal vein declamping, we will start rapid 500 ml 4% albumin infusion or packed RBCs (according to the anhepatic hemoglobin level 5 min before declamping) through 14 Gauge peripheral venous cannula in all patients.

For hypotension we will give norepinephrine and for resistant hypotension we will use adrenaline as rescue.

Technique of ONSD:

Sonographic measurement of ONSD was performed with the same manner of previous studies. Patients were placed in the supine position with their eyes closed, and a thick gel layer was applied to the closed upper eyelid. The 7.5-MHz linear probe was placed on the gel without excessive pressure and adjusted to the proper angle for displaying the entry of the optic nerve into the globe. The intensity of the ultrasound was adjusted to display optimal contrast between the retrobulbar echogenic fat tissue and the vertical hypoechoic band. An ultrasound beam was focused on the retrobulbar area using the lowest possible acoustic power that could measure ONSD. The ONSD was measured 3 mm behind the optic disc. Measurements were performed in the transverse and sagittal planes of both eyes, and the ﬁnal ONSD value was calculated by averaging 4 measured values. (8)

Immunosuppression:

All patients will receive intravenous 0.5 gm methylprednisolone at the start of the warm ischemia. After hepatic artery anastomosis and declamping, we will administer 500 mg mycophenolate mofetil through the nasogastric tube and i.v. 20 mg basiliximab.

In the ICU, patients will receive oral tacrolimus starting the day after the operation (adjusting the dose targeting serum level of 5-10 ng/ml) , mycophenolate mofetil 500 mg twice per day and basiliximab 20 mg iv 4 days after.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients of both sex undergoing living donor liver transplantation operation

Exclusion Criteria:

* History of optic neuritis
* History of Arachnoid cyst of the optic nerve.
* History of eye trauma
* History of optic nerve trauma.
* Familial amylodotic polyneuropathy
* Wilson disease.
* Patient planned to use immunosuppression regimen other than tacrolimus.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult (>= 18 years) recipients undergoing living donor liver transplantation
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-03-23 (Actual); Study Completion 2021-03-23 (Actual)

PRIMARY OUTCOMES:
Early tacrolimus neurotoxicity | 28 days after transplantation
  definition that will be considered when neurological events (visual disturbance, altered level of consciousness, confusion, psychosis, seizure, encephalopathy, tremors and/or coma or change in the pattern of the preexisting cirrhotic neurological changes ) appeared in the absence of central pontine myelinolysis, central nervous system infection, stroke, or hemorrhage within the first 4 weeks after LT and symptoms improved after dose modification of CNI therapy

SECONDARY OUTCOMES:
Time and presentation of neurotoxicity | 28 days after transplantation
  according to the 1ry outcome definition, the time (day) and presentation (clinically) reported
Intensive Care Unit stay | until discharge from ICU for 1 year
  reported in days
Hospital Length of stay | until discharge from the hospital for 1 year
  Measured in days
Mortality | three months after transplant
  three-month all-cause mortality

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud M. Elsedeiq, MD, Principal Investigator — Lecturer of anaesthesia and intensive care; Amr M. Yassin, MD, Study Director — professor of anaesthesia and surgical intensive care
Locations (1):
- Gastroenerology Surgical Center - Liver transplantation program, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Elsedeiq M, Abdelkhalek M, Abozeid KM, Habl MS, Elmorshedi MA, Yassen AM, Emara MM. Intraoperative Optic Nerve Sheath Diameter as a Predictor of Early Tacrolimus Neurotoxicity after Living Donor Liver Transplantation. Anaesth Crit Care Pain Med. 2023 Feb;42(1):101178. doi: 10.1016/j.accpm.2022.101178. Epub 2022 Nov 25. PMID 36442803